CLINICAL TRIAL: NCT04973423
Title: STUDY OF THE ADDED VALUE OF A TRANSMURAL EVALUATION IN PATIENTS WITH CROHN'S DISEASE UNDER BIOTHERAPY WITH CLOSE FECAL CALPROTECTIN FOLLOW-UP
Acronym: Deeper
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHRC IR 2020 BUISSON
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Crohn Disease; Calprotectin; MRI
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CALM (No Intervention): Tight control of inflammatory activity by calprotectin.
- CALM + IRM (Other): Tight control of inflammatory activity by calprotectin associated with transmural evaluation.
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — 2 additional MRI will be done for the CALM + MRI group
  Arms: CALM + IRM

SUMMARY:
Crohn's disease (CD) is a chronic inflammatory bowel disease (IBD) that can dramatically affect the quality of life of patients. Due to its transmural nature (involvement of the entire thickness of the intestinal wall), it naturally progresses to intestinal destruction (stenosis, fistula) which requires intestinal resection in approximately half of patients during their follow-up. The long-term goal for patients is to maintain a normal life, that is, without symptoms and without intestinal destruction. For this, the short and medium term therapeutic objectives have evolved in recent years. Clinical remission is not a sufficient goal since it has failed to alter the natural history of the disease. The current objective to be achieved is the combination of clinical remission and endoscopic mucosal healing since it is associated with a reduced risk of progression (reappearance of symptoms, hospitalization, intestinal resection). Fecal calprotectin, better accepted than colonoscopy, is a non-invasive biomarker of endoscopic inflammatory activity in CD. The CALM study recently showed that close follow-up with clinical and biological evaluation (assays of CRP and fecal calprotectin), called "tight control", associated with therapeutic intensification in the absence of clinical or biological remission, was associated with a better rate of endoscopic mucosal healing at 1 year than follow-up based solely on symptoms. Thus, the "CALM" strategy is considered to be the current benchmark.

Transmural healing evaluated by MRI is also a promising objective associated with a reduced risk of progression (reappearance of symptoms, hospitalization, bowel resection). In addition, it could prevent intestinal destruction. A recent study by our team suggested that calprotectin (mucosal assessment) and MRI (transmural assessment) may be complementary and be a better therapeutic goal. We hypothesize that a "CALM + MRI" strategy concomitantly targeting transmural healing would be superior to the "CALM" strategy alone in maintaining clinical remission without corticosteroids in patients with CD treated with biotherapies.

DETAILED DESCRIPTION:
This is a randomized, open-label controlled study comparing two therapeutic strategies in patients with CD (see inclusion criteria) starting biotherapy. Randomization, by minimization (Stata version 15), will be stratified by center, by biotherapy line and on the location of the disease: MC colic isolated (L2 according to the Montreal classification) vs. Ileal or ileocolic MC (L1 + L3), for a maximum of L1 + L3 patients of 70%.

The reference arm will be based on that of the CALM study, i.e. regular follow-up (S0, S12, S24, S52, S76, S100, S124 and S152) with therapeutic intensification in the absence of at least one criterion among CDAI <150, CRP <5 or fecal calprotectin <250. After checking the inclusion criteria, the patients will be included and randomized. The initial choice of biotherapy, therapeutic intensifications (dose increase, interval reduction, treatment change) and treatment sequences will be based on the French consensus of 2020. MRI will be performed in all patients at weeks 0, 76 and 152. In the MRI arm, an additional MRI will be performed at W24 and W52 with therapeutic intensification at W24, W52 and W76 in the presence of residual MRI activity. Patients will be followed for 152 weeks (≈ 3 years). In the event of a missing examination (calprotectin or MRI), the intensification will be carried out or not with the available data. Therefore, the analysis will be performed by intention to treat (ITT). Patients will be given a symptom calendar (abdominal pain score (between 0 = no pain and 3 = severe pain) and number of stools). Each month without data (lost to follow-up) will be considered as in the absence of clinical remission without corticosteroids (ITT). The fecal calprotectin dosage will be standardized and performed with the same test in all patients. Therapeutic intensification based on MRI will be carried out after a centralized review. The secondary endpoints (response and transmural healing, Lémann index) will be centrally blinded in the study arm to avoid any evaluation bias.

ELIGIBILITY:
Inclusion Criteria:

* Adult Crohn's disease (age ≥ 18 years)
* Symptomatic with Crohn's disease activity index (CDAI)> 150
* Presence of objective signs of inflammatory activity (fecal calprotectin> 250 AND sign of MRI activity)
* Requiring treatment with biotherapy according to the investigator
* Able to give informed consent to participate in research
* Affiliation to a Social Security scheme.

Exclusion Criteria:

* Severe obstructive symptoms
* Uncontrolled intra-abdominal abscess
* Isolated anoperineal lesions
* Prevention of postoperative endoscopic recurrence
* Temporary or definitive ostomy
* Total colectomy
* Contraindication to MRI
* Pregnant or breastfeeding women
* Protected adults (curatorship, guardianship, saving justice)
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2027-03-21 (Estimated); Study Completion 2027-08-21 (Estimated)

PRIMARY OUTCOMES:
Proportion of months spent in clinical remission | Between week 24 and week 76.
  Proportion of months (4 week period) spent in clinical remission without corticosteroids according to PRO-2 (<3 very soft or watery stools per day and no moderate to severe abdominal pain).

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Amiens university hospital, Amiens
  - Aurillac Hospital, Aurillac
  - Bayonne hospital, Bayonne
  - Bordeaux university hospital, Bordeaux
  - Chambery Hospital, Chambéry
  - Clermont-Ferrand University hospital, Clermont-Ferrand
  - Grenoble University Hospital, Grenoble
  - Issoire Hospital, Issoire
  - LILLE university hospital, Lille
  - Lyon Hospital, Hospices civils de Lyon, Lyon
  - Montluçon Hospital, Montluçon
  - Montpellier University hospital, Montpellier
  - Nancy University hospital, Nancy
  - Nice University hospital, Nice
  - Rennes University Hospital, Rennes
  - Saint Etienne University Hospital, Saint-Etienne
  - Thiers Hospital, Thiers